CLINICAL TRIAL: NCT04814290
Title: Long-term Follow-up of Living Liver Donors: A Single-center Experience
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Shehta, MD, PhD, Mansoura University
Other Study IDs: No. MD/15.08.50
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Liver Transplantation
Keywords: Living-donor liver transplantation; Quality of life; Follow up
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- living liver donors: cases already underwent hepatectomy for living-donor liver transplantation.
  Interventions: Other: health-related quality of life (HRQoL) (36-item short-form health survey, version 1 [SF-36]).
- matched controls: healthy persons who attended the preoperative clinic while preparing for donation but were rejected because of an ABO blood group mismatch.
  Interventions: Other: health-related quality of life (HRQoL) (36-item short-form health survey, version 1 [SF-36]).

INTERVENTIONS:
Other: health-related quality of life (HRQoL) (36-item short-form health survey, version 1 [SF-36]). — health-related quality of life (HRQoL) (36-item short-form health survey, version 1 [SF-36]).

SUMMARY:
Data on the long-term consequences of living liver donation are scarce. This study examined clinical, laboratory, and radiological parameters and long-term health-related quality of life (HRQoL) in 237 living liver donors and 239 matched controls during 48 to 168 months of postdonation follow-up.

DETAILED DESCRIPTION:
Data on the long-term consequences of living liver donation are scarce. This study examined clinical, laboratory, and radiological parameters and long-term health-related quality of life (HRQoL) in 237 living liver donors and 239 matched controls during 48 to 168 months of postdonation follow-up.

We used the 36-item short-form health survey (short form-36 health survey, version 1 [SF-36]). The scores for the 4 following subscales were higher in nondonors than in donors: physical functioning (P = 0.009), role limitations due to physical health (P = 0.002), energy/fatigue (P < 0.001), and bodily pain (P < 0.001). The scores on the 8 subscales of the SF-36 were higher in donors with living recipients than in donors whose recipients died (P < 0.001). Our results suggest that living donor right hepatectomy is safe and results in a postdonation HRQoL similar to that of nondonors in those donors whose recipients are healthy, while donors whose recipients die have a lower HRQoL that is significantly negatively correlated with the time since recipient death and improves over time.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years
* no comorbidities.
* BMI less than 30 kg/m2.
* compatible ABO group.

Exclusion Criteria:

* Older than 50 years.
* Associated comorbidities.
* Obesity.
* Noncompatible ABO group.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: 237 living liver donors and 239 matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2004-05-01 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
health-related quality of life (HRQoL) | 4 to 16 years of follow up
  health-related quality of life (HRQoL) (36-item short-form health survey, version 1 [SF-36]).

IPD SHARING:
Plan to Share IPD: Undecided
Privacy for liver transplantation unit, mansoura university.